CLINICAL TRIAL: NCT06397326
Title: Sustainable and Healthy Return-to-Work Program for Employees of Large Healthcare Organizations - PRATICAdr 2.0
Brief Title: Sustainable and Healthy Return-to-Work Program - PRATICAdr 2.0
Acronym: PRATICAdr
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec a Montréal (Other)
Collaborators: Centre intégré de santé et de services sociaux (CISSS) de la Gaspésie (Unknown); Centre intégré de santé et de services sociaux (CISSS) de Laval (Unknown); Centre hospitalier de l'Université de Montréal (CHUM) (Other); Centre intégré universitaire de santé et de services sociaux du Centre Ouest de Montréal (Unknown)
Responsible Party: Principal Investigator, Marc Corbière, Full professor, Université du Québec a Montréal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MSSS-23-RH-00599
Record Dates: First submitted 2024-04-05; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Common Mental Disorder
Keywords: Return to work; Sick leave duration; Relapses; Clinical symptoms
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Intervention Model Description: Two groups:
  Experimental: Return to work coordinator + PRATICAdr 2.0 Control group: Return to work coordinator only
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Return to work coordinator + PRATICAdr 2.0 (Experimental): The primary objective of the Return to work coordinator (RTW-C) is to coordinate, plan, and promote sustainable RTW for employees on sick leave.The RTW-C is responsible for assessing employee functioning while exploring barriers to RTW and available resources to develop a RTW plan. Also, RTW-C enhance communication and collaboration among stakeholders involved in the RTW process.
  In this arm, the RTW-C uses PRATICAdr 2.0, a web application including key features (e.g., Facilitation of collaboration among multiple RTW stakeholders across healthcare, enterprise, and insurance sectors; Integration of each stakeholder's action into the sick leave employee's RTW process; sequential process aligned with the three phases of the RTW, inclusion of tools).
  Interventions: Behavioral: Return to work coordinator + PRATICAdr 2.0
- Return to work coordinator only (Sham Comparator): The primary objective of the Return to work coordinator (RTW-C) is to coordinate, plan, and promote sustainable RTW for employees on sick leave.The RTW-C is responsible for assessing employee functioning while exploring barriers to RTW and available resources to develop a RTW plan. Also, RTW-C enhance communication and collaboration among stakeholders involved in the RTW process.
  In this arm, the RTW-C does not use PRATICAdr 2.0.
  Interventions: Behavioral: Return to work coordinator only

INTERVENTIONS:
Behavioral: Return to work coordinator + PRATICAdr 2.0 — The Return to work coordinator (RTW-C) uses PRATICAdr. 2.0 (web application).
  Arms: Return to work coordinator + PRATICAdr 2.0
Behavioral: Return to work coordinator only — The Return to work coordinator (RTW-C) intervenes on employees on sick leave as usual
  Arms: Return to work coordinator only

SUMMARY:
This study aims to assess the effectiveness of PRATICAdr 2.0, a web application facilitated by a Return-to-Work Coordinator (RTW-C), with a focus on reducing sick leave duration and preventing relapse in individuals with CMDs. PRATICAdr 2.0 designed to enhance collaboration among Return-to-Work (RTW) stakeholders and provide systematic support throughout the RTW process, is evaluated in a randomized control trial (RCT). As part of the RCT, a total of 80 sick leave employees from 4 large public health organizations (n=80, 40 from the experimental group and 40 from the control group) will be recruited. The control group receives usual services offered by a RTW-C to sick leave employees, while the experimental group receives RTW-C services plus the use of PRATICAdr 2.0.

DETAILED DESCRIPTION:
Common mental disorders (CMDs) are highly prevalent in workplace settings, and have become a significant public health challenge. This study aims to assess the effectiveness of PRATICAdr 2.0, a web application facilitated by a Return-to-Work Coordinator (RTW-C), with a focus on reducing sick leave duration and preventing relapse in individuals with CMDs. PRATICAdr 2.0 designed to enhance collaboration among Return-to-Work (RTW) stakeholders and provide systematic support throughout the RTW process, is evaluated in a randomized control trial (RCT). As part of the RCT, a total of 80 sick leave employees from 4 large public health organizations (n=80, 40 from the experimental group and 40 from the control group) will be recruited. The control group receives usual services offered by a RTW-C to sick leave employees, while the experimental group receives RTW-C services plus the use of PRATICAdr 2.0. Participants will be randomly assigned to either the PRATICAdr 2.0 experimental group or the control group using computerized stratified randomization based on age, site, and sex (sealed envelope method). Participants will complete a series of online questionnaires at several following time points. Survival analyses were used to compare sick leave durations and relapses between the experimental group (PRATICAdr with RTW-C), and control groups (RTW-C only). Mixed linear models were used to observe changes in clinical symptoms over time, especially for the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Sick leave due to Common mental disorder (i.e. depression, anxiety, adjustment disorder, burnout)
* Sick leave duration (from 1 to 3 months)
* Member of participating unions in the large health organization

Exclusion Criteria:

* Inability to communicate in French
* Have a known organic disorder
* Have a professional dirsorder (CNESST)
* Have experienced previous sick leaves due to Common mental disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Sick leave duration | through study completion, an average of 2 years
  The number of days during the sick leave
Relapses | through study completion, an average of 2 years
  Number of relapses after returning to work

SECONDARY OUTCOMES:
Depressive symptoms | through study completion, an average of 2 years
  Patient Health Questionnaire for depression (PHQ-9; Kroenke et al., 2001)
Anxiety symptoms | through study completion, an average of 2 years
  Generalized Anxiety Disorder Scale (GAD-7; Spitzer et al., 2006)
Return to Work Obstacles and Self-Efficacy | through study completion, an average of 2 years
  Return to Work Obstacles and Self-Efficacy Scale (ROSES ; Corbière et al., 2017 )

OTHER OUTCOMES:
Social functioning | through study completion, an average of 2 years
  WHODAS
Working alliance | through study completion, an average of 2 years
  Working Alliance Inventory (Horvath & Greenberg, 1989; Corbière et al., 2006)
Work accommodations | through study completion, an average of 2 years
  Work Accommodation and Natural Support Scale (WANSS; Corbière et al., 2014)
Work recognition | through study completion, an average of 2 years
  Recognition by stakeholders of returning to work following a common mental disorder (RECONNECT, Corbière, Larivière, Charette-Dussault, 2021)